CLINICAL TRIAL: NCT03424395
Title: A Clinical Trial to Evaluate the Effects of Proprietary Personalized Dietary Programs on Markers of Health and Wellness, Body Composition, and Quality of Life
Brief Title: Personalized Dietary Program and Markers of Wellness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Habit, LLC (Industry)
Collaborators: TNO (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Habit-1701
Record Dates: First submitted 2018-01-25; First posted 2018-02-07 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Healthy; Metabolism
Keywords: personalized dietary and wellness program; oral protein glucose lipid tolerance test; metabolism; behavior; health; body composition; single nucleotide polymorphisms; genotype; dietary and wellness coaching/advice; liquid meal challenge test
MeSH Terms: conditions — Behavior | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: Single arm (open-label) containing three periods: (1) run-in (control), (2) personalized advice/counseling and meals, (3) personalized advice/counseling only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized dietary and wellness program (Other): An integrated personalized nutrition program which includes a combination of dietary and wellness advice/counseling on wellness and meals, or dietary and wellness advice/counseling alone, each for 10 weeks.
  Interventions: Other: Personalized dietary and wellness program

INTERVENTIONS:
Other: Personalized dietary and wellness program — Single arm intervention containing three periods: (1) run-in (control), (2) personalized advice/counseling and meals, (3) personalized advice/counseling only

SUMMARY:
The objective of this study is to determine the impact of an integrated personalized dietary and wellness program which includes dietary advice, meals, and counseling on health and wellness.

DETAILED DESCRIPTION:
The objective of this study is to determine the impact of an integrated personalized dietary and wellness program, which includes personalized dietary advice, meals, and behavior guidance, on markers of health and wellness, body composition, and psychosocial measures. Behavior questionnaires, motivational interviewing, psychosocial questionnaires, and participants' self-generated data on diet, preferences, activity, and sleep will be used in combination with anthropometric and biological data (fasted blood-based measures following an oral protein glucose lipid tolerance test [liquid meal challenge test], and selected single nucleotide polymorphisms) to create individualized, tailored dietary advice, meal and counseling plans.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 30-65 years of age, inclusive.
* BMI 18.5-39.9 kilograms per meters squared.
* Willing to follow study program instructions, including consumption of meals on site (5 days/week; breakfast and lunch), consumption of all provided meals, use of a Fitbit®, self-administered capillary blood draws and dried blood spot collection, and visit schedule, where relevant.
* Willing and able to comply with the visit/contact schedule.
* Willing to avoid vigorous activity and alcohol consumption (24 h) and willing to fast (10-14 h, water only) prior to completion of the at-home oral protein glucose lipid tolerance test.
* Normally active and judged to be in good health on the basis of the medical history.
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigators.
* Subject has access to an internet-ready device and email.

Exclusion Criteria:

* A history or presence of clinically important endocrine, cardiovascular, pulmonary, hepatic, renal, hematologic, immunologic, dermatologic, neurologic, psychiatric or biliary disorders that could interfere with the interpretation of the study results.
* A history or presence of a gastrointestinal condition that could potentially interfere with digestion and absorption of the study product including, inflammatory bowel disease, irritable bowel syndrome, chronic constipation, and history of frequent diarrhea; and gastroparesis.
* Uncontrolled hypertension (systolic blood pressure ≥160 mm Hg or diastolic blood pressure ≥100 mm Hg).
* A history or presence of cancer in the prior 2 years, except for non-melanoma skin cancer.
* A history of unconventional sleep patterns.
* Major trauma or a surgical event within 3 months of screening.
* Nicotine users.
* Use of medications which can alter the lipid profile with the exception of stable statin use.
* Unstable use of any thyroid medication.
* Use of antibiotics, hypoglycemic medications, and/or systemic corticosteroids.
* Signs or symptoms of an active infection.
* Current or recent history of drug or alcohol abuse.
* Known allergy and/or sensitivity to the study foods or products.
* Extreme dietary habits (e.g., very high protein diets, vegan, very low carbohydrate, etc.).
* A change (increase or decrease) in body weight of >10%.
* Females who are pregnant, planning to be pregnant during the study period, lactating, or of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
* Study staff or those who will be involved in the conduct of the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-10-28 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change in metabolic composite score | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  A composite score that includes aggregated changes in blood biomarkers (glucose, C-peptide, high-density lipoprotein cholesterol, total cholesterol, and triglyceride levels).

SECONDARY OUTCOMES:
Change in blood pressure | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  systolic and diastolic blood pressures
Change in body mass index | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in quality of life | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  composite score and individual ratings from the WHOQOL-BREF questionnaire
Change in sleep time | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  weekly averages of hours from a Fitbit®
Change in ratings of diet/food behavior | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  composite score from the Diet Self-efficacy Questionnaire and Food Behavior and Activity Inventory
Change in activity | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  weekly averages of hours from a Fitbit®
Change in food intake | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  weekly averages of nutrients and food intake from diet records
Change in heart rate | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in body weight | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in waist circumference | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in hip circumference | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in fat-free mass | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in fat mass | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
Change in stress | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  composite score and individual ratings from the Perceived Stress Scale
Change in C-peptide | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  The change from 0 to 30 min, 0 to 120 min, and area under the curve from 0 to 120 min pre- and post-oral protein glucose lipid tolerance test (liquid meal challenge test).
Change in disposition index | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  The change from 0 to 30 min, 0 to 120 min, and area under the curve from 0 to 120 min pre- and post-oral protein glucose lipid tolerance test (liquid meal challenge test).
Changes in insulin indices | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  The change from 0 to 30 min, 0 to 120 min, and area under the curve from 0 to 120 min pre- and post-oral protein glucose lipid tolerance test (liquid meal challenge test) for hepatic insulin index and Matsuda insulin sensitivity index.
Changes in lipid paramaters | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  The change from 0 to 30 min, 0 to 120 min, and area under the curve from 0 to 120 min pre- and post-oral protein glucose lipid tolerance test (liquid meal challenge test) for total cholesterol, low-density lipoprotein cholesterol, high-density lipoprotein cholesterol, and triglycerides.
Change in glucose | The change between the run-in (control) period (baseline; 10 weeks) and each intervention period (personalized advice + meals or personalized advice only; 10 weeks each)
  The change from 0 to 30 min, 0 to 120 min, and area under the curve from 0 to 120 min pre- and post-oral protein glucose lipid tolerance test (liquid meal challenge test).

CONTACTS AND LOCATIONS:
Overall Officials: Joshua C Anthony, PhD, Principal Investigator — Habit, LLC; Barbara L Winters, PhD, RD, Principal Investigator — Winters Nutrition Associates LLC; Kristin M Nieman, PhD, Study Director — Katalyses LLC
Locations (1):
- Campbell Soup Company, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Blaak EE, Hul G, Verdich C, Stich V, Martinez A, Petersen M, Feskens EF, Patel K, Oppert JM, Barbe P, Toubro S, Anderson I, Polak J, Astrup A, Macdonald IA, Langin D, Holst C, Sorensen TI, Saris WH. Fat oxidation before and after a high fat load in the obese insulin-resistant state. J Clin Endocrinol Metab. 2006 Apr;91(4):1462-9. doi: 10.1210/jc.2005-1598. Epub 2006 Jan 31. PMID 16449343
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Friedewald WT, Levy RI, Fredrickson DS. Estimation of the concentration of low-density lipoprotein cholesterol in plasma, without use of the preparative ultracentrifuge. Clin Chem. 1972 Jun;18(6):499-502. No abstract available. PMID 4337382
- [Background] Hardcastle SJ, Taylor AH, Bailey MP, Harley RA, Hagger MS. Effectiveness of a motivational interviewing intervention on weight loss, physical activity and cardiovascular disease risk factors: a randomised controlled trial with a 12-month post-intervention follow-up. Int J Behav Nutr Phys Act. 2013 Mar 28;10:40. doi: 10.1186/1479-5868-10-40. PMID 23537492
- [Background] Horne JA, Ostberg O. A self-assessment questionnaire to determine morningness-eveningness in human circadian rhythms. Int J Chronobiol. 1976;4(2):97-110. PMID 1027738
- [Background] Hunot C, Fildes A, Croker H, Llewellyn CH, Wardle J, Beeken RJ. Appetitive traits and relationships with BMI in adults: Development of the Adult Eating Behaviour Questionnaire. Appetite. 2016 Oct 1;105:356-63. doi: 10.1016/j.appet.2016.05.024. Epub 2016 May 20. PMID 27215837
- [Background] Johnson RK. Dietary intake--how do we measure what people are really eating? Obes Res. 2002 Nov;10 Suppl 1:63S-68S. doi: 10.1038/oby.2002.192. No abstract available. PMID 12446861
- [Background] Kardinaal AF, van Erk MJ, Dutman AE, Stroeve JH, van de Steeg E, Bijlsma S, Kooistra T, van Ommen B, Wopereis S. Quantifying phenotypic flexibility as the response to a high-fat challenge test in different states of metabolic health. FASEB J. 2015 Nov;29(11):4600-13. doi: 10.1096/fj.14-269852. Epub 2015 Jul 21. PMID 26198450
- [Background] Kolodziejczyk JK, Norman GJ, Roesch SC, Rock CL, Arredondo EM, Madanat H, Patrick K. Exploratory and confirmatory factor analyses and demographic correlate models of the strategies for weight management measure for overweight or obese adults. Am J Health Promot. 2015 Mar-Apr;29(4):e147-57. doi: 10.4278/ajhp.130731-QUAN-391. Epub 2014 Mar 26. PMID 24670075
- [Background] Kristal AR, Kolar AS, Fisher JL, Plascak JJ, Stumbo PJ, Weiss R, Paskett ED. Evaluation of web-based, self-administered, graphical food frequency questionnaire. J Acad Nutr Diet. 2014 Apr;114(4):613-21. doi: 10.1016/j.jand.2013.11.017. Epub 2014 Jan 24. PMID 24462267
- [Background] Resnicow K, McMaster F. Motivational Interviewing: moving from why to how with autonomy support. Int J Behav Nutr Phys Act. 2012 Mar 2;9:19. doi: 10.1186/1479-5868-9-19. PMID 22385702
- [Background] Stewart EE, Fox CH. Encouraging patients to change unhealthy behaviors with motivational interviewing. Fam Pract Manag. 2011 May-Jun;18(3):21-5. No abstract available. PMID 21842805
- [Background] Stich C, Knauper B, Tint A. A scenario-based dieting self-efficacy scale: the DIET-SE. Assessment. 2009 Mar;16(1):16-30. doi: 10.1177/1073191108322000. Epub 2008 Aug 14. PMID 18703821
- [Background] Stroeve JHM, van Wietmarschen H, Kremer BHA, van Ommen B, Wopereis S. Phenotypic flexibility as a measure of health: the optimal nutritional stress response test. Genes Nutr. 2015 May;10(3):13. doi: 10.1007/s12263-015-0459-1. Epub 2015 Apr 21. PMID 25896408
- [Background] Teeter BS, Kavookjian J. Telephone-based motivational interviewing for medication adherence: a systematic review. Transl Behav Med. 2014 Dec;4(4):372-81. doi: 10.1007/s13142-014-0270-3. PMID 25584086
- [Background] van Amelsvoort JM, van Stratum P, Kraal JH, Lussenburg RN, Houtsmuller UM. Effects of varying the carbohydrate:fat ratio in a hot lunch on postprandial variables in male volunteers. Br J Nutr. 1989 Mar;61(2):267-83. doi: 10.1079/bjn19890115. PMID 2650734
- [Background] van Ommen B, van der Greef J, Ordovas JM, Daniel H. Phenotypic flexibility as key factor in the human nutrition and health relationship. Genes Nutr. 2014 Sep;9(5):423. doi: 10.1007/s12263-014-0423-5. Epub 2014 Aug 9. PMID 25106484
- [Background] Development of the World Health Organization WHOQOL-BREF quality of life assessment. The WHOQOL Group. Psychol Med. 1998 May;28(3):551-8. doi: 10.1017/s0033291798006667. PMID 9626712
- See also: Institute of Medicine - Dietary Reference Intakes — http://doi.org/10.17226/10490
- See also: World Health Organization - Physical Activity Definitions — http://www.who.int/dietphysicalactivity/physical_activity_intensity/en/
- See also: World Health Organization: Waist and Hip Circumference Ratio — http://apps.who.int/iris/bitstream/10665/44583/1/9789241501491_eng.pdf